CLINICAL TRIAL: NCT01708928
Title: Feasibility Study: Evaluation Of The Ulthera™ System For Obtaining Lift And Tightening Of The Neck Skin In Patients With A History Of Submentoplasty And Or Rhytidectomy Vs Patients Naïve To Submentoplasty Or Rhytidectomy - A Feasibility Study
Brief Title: Feasibility Study: Lifting and Tightening Neck Skin in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-107
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Subjects who have previous history of submentoplasty and or rhytidectomy
  Interventions: Device: Ulthera System Treatment
- Group B (Active Comparator): Subjects naïve to submentoplasty and or rhytidectomy
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 30 subjects will be enrolled. All subjects will receive one Ultherapy treatment to the lower two thirds of the face and neck. Subjects will be equally grouped into those with a history of submentoplasty and or rhytidectomy and those naive to submentoplasty and or rhytidectomy. Follow-up visits will occur at 14, 30, 60, 90 and 180 days following treatment. Study images will be obtained pre-treatment, 30-60 minutes post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective single center study. Subjects will be enrolled one per group as they present. Efficacy will be determined by the change in submental volume and cervicomental angle. GAIS and patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years
* Subject in good health
* Body Mass index of less than 30
* Present with unwanted skin laxity in the submental area as demonstrated by a grade 2 or 3 on the Knize scale for classification of cosmetic deformity of the cervicomental angle
* Previous history of surgical submentoplasty and or rhytidectomy greater than 12 months previous to enrollment and not to exceed 120 months prior to enrollment
* Understands and accepts the obligation not to receive any other procedures in the submental areas thru the 6 month follow up visit
* Willingness and ability to comply with protocol requirements including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study
* Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control

Exclusion Criteria:

* Pregnant, lactating or planning to become pregnant and or not using a reliable form of birth control
* Has an active systemic or local skin disease that may alter wound healing
* Subjects with a prior cosmetic or medical history of submentoplasty and or Rhytidectomy within the last 12 months or greater than 120 months
* Subjects with a prior cosmetic or medical history of submentoplasty and or Rhytidectomy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in submental volume | 90 days post-treatment
  Measured by the Canfield Vectra® imaging system comparing pre-treatment baseline photos to post-treatment photos.

SECONDARY OUTCOMES:
Overall improvement of the submental area | 90 days post-treatment
  Global Aesthetic Improvement Scale (GAIS) and patient satisfaction questionnaires will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States